CLINICAL TRIAL: NCT06255171
Title: Social Media and Suicidal Behaviour: a Study of the Impact of Suicide Related Journalistic Publications on Commentators and Readers - Study 1
Brief Title: Social Media and Suicidal Behaviour - Study 1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J3-3081-1
Record Dates: First submitted 2024-01-17; First posted 2024-02-13 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Suicidal Behaviour
Keywords: social media; suicide; reporting on suicide; university students; impact of reporting; suicidal behaviour
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to one of 3 arms, one of which will be an experimental group and 2 will be control groups.
Who Masked: Participant
Masking Description: Participants will know that they are allocated to one of 3 arms, but will not know if the arm is a control group or experimental. After the main part of the study, all groups of participants will be involved in a group debriefing conversation, providing an opportunity for feedback from both the study's facilitators and participants. It will facilitate clarification of conditions (experimental or control group) and provide a platform for discussing participants' feelings, potential dilemmas, questions, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nature articles - control 1 (Other): Participants will read posts and articles about nature.
  Interventions: Behavioral: Reading journalistic posts and articles on social media on nature
- Death by suicide articles (Experimental): Participants will read posts and articles about death by suicide.
  Interventions: Behavioral: Reading journalistic posts and articles on social media on deaths by suicide
- Articles about traffic-related deaths - control 2 (Other): Participants will read posts and articles about traffic-related deaths.
  Interventions: Behavioral: Reading journalistic posts and articles on social media on traffic-related deaths

INTERVENTIONS:
Behavioral: Reading journalistic posts and articles on social media on nature — Reading journalistic posts and articles, published on social media, regarding nature.
  Arms: Nature articles - control 1
Behavioral: Reading journalistic posts and articles on social media on deaths by suicide — Reading journalistic posts and articles, published on social media, regarding deaths by suicide.
  Arms: Death by suicide articles
Behavioral: Reading journalistic posts and articles on social media on traffic-related deaths — Reading journalistic posts and articles, published on social media, regarding traffic-related deaths
  Arms: Articles about traffic-related deaths - control 2

SUMMARY:
There is limited research investigating the correlation between suicidal behavior in the general population and online journalism reporting on suicide. Even less explored are the roles and characteristics of suicide-related news posts on social media platforms, along with reader comments, and their association with users' experiences. The primary objective of this randomized controlled trial is to experimentally examine the influence of these post features on user perceptions. Participants are expected to be university students or young adults.

In line with this aim, the following research question has been posed:

How do users of social media and forums perceive news posts about suicide on social media platforms?

Participants will complete a screening battery of questionnaires. Those who will be eligible to participate will be divided into 1 experimental and 2 control groups. Firstly the participants will fill out a questionnaire regarding their current mood. Each group will read posts of a different theme, one of them will be suicidal behavior, deaths due to traffic accidents, and nature. They will be asked to observe and read 4 social media posts and their corresponding articles. After each article, they will answer a few questions on how they perceived these articles and how are they currently feeling. After the main part of the study, all groups of participants will be involved in a group debriefing conversation.

DETAILED DESCRIPTION:
The clinical trial will comprise three samples:

* The experimental group sample (experimental condition: reading articles on death by suicide). Experimental group sample will include 20-25 adult residents of Slovenia.
* The first control group sample (control condition: reading articles on deaths due to traffic accidents). First control group sample will include 20-25 adult residents of Slovenia.
* The second control group sample (control condition: reading neutral articles about nature). Second control group sample will include 20-25 adult residents of Slovenia.

The total number of participants in all three groups will range from 60 to 80 individuals, they will be recruited through various channels. The research group will disseminate the link to the online invitation using the 1KA platform, along with a request for its dissemination to the departments of the University of Primorska and other public universities in Slovenia. Members of the research team will also share the research invitation with their students. Recruitment will be extended through media announcements, our website zivziv.si, and our Facebook account, UP Insititute Andrej Marušič. Additional invitations to participate in the study may be extended through brief presentations in courses across different academic disciplines, in collaboration with the respective course instructors.

The research invitation will be freely accessible online and will include information about the compensation for participation. The invitation will also include a consent form, which participants will provide at the first stage and which will cover all further stages of study participation. The online consent form will be presented on the 1KA platform.

The sample will exclusively include adult residents of Slovenia. Participants who receive the invitation and decide to participate will:

i) Read detailed instructions about the project and participation and complete an informed consent: Clicking on the link will take potential participants to the first step of research participation on the 1KA platform. They will read all the relevant information about the purpose, implementation, and then proceed to complete an informed consent indicating their conscious decision to participate. If participants provide all necessary information and the informed consent for participation, they will receive a link to the next step on the 1KA platform-completing a battery of questionnaires for screening purposes (detailed in the section on the description of methods).

ii) Complete the screening battery of questionnaires: Participants will then receive a link to a battery of questionnaires assessing subjective well-being, the presence of depression symptoms, and/or suicidal thoughts. After completing the questionnaire battery on the 1KA platform, all participants will receive an invitation to participate in the experimental laboratory study or a notice of potential rejection via their provided email address. The rejection notice will include an explanation of the rejection, sources of assistance in distress, the significance of seeking help, and our contact information. This notice will be sent to those participants who exhibit diminished subjective well-being, the presence of depression symptoms, and/or suicidal thoughts for their safety and well-being, excluding them from the study.

Participants who do not exceed the predefined threshold values will be invited to participate in the main part of the study.

iii) Participate in the main part of the study (experimental and control groups): The main part of the study will include the experimental group and two control groups of participants. Participants will be randomly assigned to groups, ensuring that the experimental and control groups are comparable in terms of the number of participants, gender, age, and their field of study or achieved education level (social sciences or natural sciences). Other characteristics of participants cannot be predicted at this stage.

Participants will receive instructions for participating in the study. Potential participants will be informed that the remainder of the study will involve in-person participation under various experimental conditions (exposure to one of three different content modules). Each participant will be exposed to only one condition and its corresponding content module, but they will not know which one before or during active participation in the study. Participants will be informed in advance that they will not know which condition they are randomly assigned to during the exposure. This approach aims to ensure transparency while achieving valid findings. Participants will be informed of their assigned condition immediately after completing their participation in the main part of the study. After the main part of the study, all groups of participants will be involved in a group debriefing conversation, providing an opportunity for feedback from both the study's facilitators and participants. It will facilitate clarification of conditions (experimental or control group) and provide a platform for discussing participants' feelings, potential dilemmas, questions, etc.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* providing an informed consent for participation in the study
* not exceeding the limit values on any of the questionnaires of the screening battery

Exclusion Criteria:

* under the age of 18
* not providing an informed consent for participation in the study
* exceeding the limit values on at least one questionnaire of the screening battery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The experience of a social media user when reading posts | Approximately 1 minute after being presented each social media post
  For the purposes of this study, questions were formulated about the experience of publication

SECONDARY OUTCOMES:
Self-rating of mood - Pleasant-Unpleasant Scale | Before and approximately 1 minute after being presented each social media post
  Using the Brief Mood Introspection Scale; BMIS; Mayer in Gaschke, 1988. Pleasant-Unpleasant Scale, min = 16, max = 64, a higher score indicating a more pleasant mood
Self-rating of mood - Arousal-Calm Mood Scale | Before and approximately 1 minute after being presented each social media post
  Using the Brief Mood Introspection Scale; BMIS; Mayer in Gaschke, 1988. Arousal-Calm Scale, min = 12, max = 48, a higher score indicating a more aroused mood

CONTACTS AND LOCATIONS:
Overall Officials: Diego De Leo, Study Director — University of Primorska; Vita Poštuvan, Principal Investigator — University of Primorska
Locations (1):
- University of Primorska, Koper, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project description in Sicris database (en) — https://cris.cobiss.net/ecris/si/en/project/18731
- See also: Opis projekta v bazi Sicris (slo) — https://cris.cobiss.net/ecris/si/sl/project/18731

DOCUMENTS (1):
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT06255171/ICF_000.pdf